CLINICAL TRIAL: NCT01391377
Title: The Effects of Chronic High-density Lipoprotein (HDL) Elevation With Extended Release Niacin on Peripheral Arterial Disease
Brief Title: Effects of Niacin on Good Cholesterol in People With Peripheral Arterial Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Tredaptive has been suspended worldwide
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 126-11
Record Dates: First submitted 2011-04-05; First posted 2011-07-12 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Peripheral Arterial Disease
Keywords: HDL; High density Lipoprotein; Peripheral arterial disease; Tredaptive; Niacin; Laropiprant; Plaque; Atherosclerosis; Lipid content
MeSH Terms: conditions — Peripheral Arterial Disease; Plaque, Amyloid; Atherosclerosis | interventions — Niacin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niacin / Laropiprant (Active Comparator)
  Interventions: Drug: Niacin/Laropiprant combination
- Sugar Pill (Placebo) (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Niacin/Laropiprant combination — Niacin 1g / Laropiprant 20mg for 4 weeks followed by Niacin 2g / Laropiprant 20mg for 4 weeks
  Other Names: Tredaptive
  Arms: Niacin / Laropiprant
Drug: Sugar pill — Placebo
  Other Names: Placebo
  Arms: Sugar Pill (Placebo)

SUMMARY:
Atherosclerosis is a disorder in the body that is characterized by cholesterol plaque formation in various arteries, causing narrowing of the artery and a limitation in blood flow. Depending on which artery the plaque is in, different clinical conditions occur. In adults common areas include in the heart arteries, in the neck arteries and in the aorta and lower leg arteries. When it affects the lower limbs it is known as peripheral arterial disease - PAD.

The main symptom of PAD is called "claudication" and is described as pain or discomfort in the legs when walking. The aim of PAD treatment is to improve walking distance and quality of life in those with intermittent claudication, and to decrease long term complications including illness and death.

An important controlling factor of these cholesterol plaques is a type of cholesterol called HDL (High density lipoprotein).

This study aims to look at the effect that raising HDL for a prolonged period has on blood markers of inflammation and on the cholesterol plaque composition in patients with PAD. This investigation will also have relevance to the effects of HDL elevation on plaque composition and inflammation in other areas of the body including the heart, neck and brain arteries.

Twenty (20) PAD patients with will be recruited into the study. The investigators anticipate recruitment of all 20 patients within 12 months. The 20 PAD patients all must have significant leg pains when walking, and after review by a doctor, be determined to have narrowings in the leg artery that they will plan to operate on. Patients will be randomized to either niacin (Tredaptive, 1g/day) or matching placebo for 8 weeks (prior to operation) After the 8 week period they will then go on to receive the normal interventional treatment as planned. Blood samples will be taken at enrollment and at the 8 week mark prior to surgery. The plaque that is removed at the time of operation will also be sent to the lab for analysis.

The investigators hope to show with this study that by raising the levels of HDL with extended release niacin, there are positive effects on the amount of cholesterol in the plaque, and on the markers in the blood of inflammation and thrombosis.

The hypothesis is that elevation of HDL with Niacin will have anti-atherosclerotic actions including: Lower plaque lipid content, Reduced plaque macrophage infiltration, Reduced monocyte activation, Reduced neutrophil adhesion, Inhibition of inflammation and Inhibition of thrombotic markers.

ELIGIBILITY:
Inclusion Criteria:

* age >40 years
* ankle-brachial index (ABI) of <0.9 at rest in at least one leg,
* symptom limiting intermittent claudication (unilateral or bilateral) and stable for the previous 6 months,
* superficial femoral artery disease amenable to percutaneous revascularisation,
* serum HDL <1.0 mmol/l
* a stable medication regime for at least 6 months

Exclusion Criteria:

* acute myocardial infarction or presentation with angina within 1 month of enrolment,
* serum creatinine >0.2mmol/l,
* significant co-morbidity with expected survival <6 months,
* current niacin or fibrate therapy
* unable to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Plaque composition | 8 weeks after recruitment.
  After femoral arthrectomy the excised plaque will analysed for histological studies, for lipid content, immunohistochemistry, macrophage content and size and VCAM-1 staining.

SECONDARY OUTCOMES:
Plasma Monocyte Activation | 8 weeks after recruitment
  Cd11b expression on peripheral blood monocytes will be measured as a marker of monocyte activation.
Plasma Neutrophil Adhesion to Immobilized Fibrinogen | 8 weeks after recruitment
Platelet Aggregation Assays | 8 weeks after recruitment
Plasma Thrombotic Markers | 8 weeks after recruitment
Size distribution and composition of HDL | 8 weeks after recruitment
Ex vivo cholesterol efflux | 8 weeks after recruitment
Plasma lipid parameters and inflammatory markers | 8 weeks after recruitment
  Lipid levels including total cholesterol, HDL, LDL and TGs, will be measured as well as ApoA1 protien and Plasma soluble ICAM-1 and soluble VCAM-1. TNF-A levels will also be measured and CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn Kingwell, Bsc, PhD, Principal Investigator — Baker IDI
Locations (1):
- Baker IDI Heart and diabetes research institute, Melbourne, Victoria, Australia